CLINICAL TRIAL: NCT04673227
Title: Cytometric Immunodiagnostics of Latent Tuberculosis Infection (LTBI) and the Influence of Previous BCG Vaccination - Pilot Study
Brief Title: Cytometric Immunodiagnostics of Latent Tuberculosis Infection (LTBI)
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Thomayer University Hospital (Other)
Collaborators: Charles University, Czech Republic (Other)
Responsible Party: Principal Investigator, Karolína Doležalová, M.D., M.D., Thomayer University Hospital
Other Study IDs: ThomayerH
Record Dates: First submitted 2020-12-12; First posted 2020-12-17 (Actual); Last update posted 2020-12-17 (Actual); Status verified 2020-12

CONDITIONS: LTBI; BCG Vaccination Reaction; TB
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Biospecimen Retention: Samples Without DNA — 30 ml of blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Contact with active TB/ LTBI: After a close contact with bacteriologically confirmed TB suspicion for LTBI with an evidence of previous BCG vaccination status TB confirmed with TST (TST ≥ 5 mm or BCG unvaccinated or TST ≥ 15 mm for BCG vaccinated) 20 children and adolescents 20 adults
  Interventions: Diagnostic Test: Blood draw
- Active TB group: Active TB group with positive microbial culture and pathological chest radiography or chest CT 20 children and adolescents 20 adults
  Interventions: Diagnostic Test: Blood draw
- Contact with active TB/ negative: After a close contact with bacteriologically confirmed TB no evidence of TB in TST or IGRA test for 3 months 20 children and adolescents 20 adults
  Interventions: Diagnostic Test: Blood draw

INTERVENTIONS:
Diagnostic Test: Blood draw — Blood draw and the analysis of blood in laboratory

SUMMARY:
TB-reactive immune cells will be tested in a multiparametric flow cytometry to distinguish an immune response for antigens of Mycobacterium spp. in TB disease/latent infection or a reaction after BCG vaccine.

DETAILED DESCRIPTION:
The goal of this project is the verification of current cytometric panel of detection antibodies in a wider panel of stimulative immunodominant antigens for CD4+ and CD8+ T cells in combination with adjuvants 2 in a in vitro activating test.

ELIGIBILITY:
Inclusion Criteria: active TB, contact with TB infection in previous 3 months before the study

-

Exclusion Criteria:

* HIV positive patients

Ages: 4 Years to 70 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Study of the broad spectrum of population with the history of having an active TB infection or close contact with bacteriologically approved pulmonary TB
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2020-01-02 (Actual); Primary Completion 2020-05-26 (Actual); Study Completion 2022-12-26 (Estimated)

PRIMARY OUTCOMES:
Peer-review publication of results of our study | 2 years

SECONDARY OUTCOMES:
Creation of new diagnostic tool and his comparision with existing IGRA test (QTF-GP and TST) | 2 years

CONTACTS AND LOCATIONS:
Locations (2):
- Czechia (2):
  - Faculty of Science, Prague
  - Thomayer Hospital, Prague

IPD SHARING:
Plan to Share IPD: No